CLINICAL TRIAL: NCT04687605
Title: Therapeutic Hypercapnia After Aneurysmal Subarachnoid Hemorrhage - Study for the Optimum Duration of Hypercapnia
Brief Title: Therapeutic Hypercapnia After Aneurysmal Subarachnoid Hemorrhage - Optimum Duration of Hypercapnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Dr. Stetter, Principial Investigator, University of Wuerzburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ230/14
Record Dates: First submitted 2020-12-22; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Vasospasm Intracranial
Keywords: SAH; Hypercapnia; DCI
MeSH Terms: conditions — Vasospasm, Intracranial; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optimum duration of hypercapnia (Experimental): Daily serial measurement of 2 hours under target hypercapnia of pCO2 50 - 55 mmHg by changes of respirator settings once per day
  Interventions: Procedure: Temporary hypercapnia

INTERVENTIONS:
Procedure: Temporary hypercapnia — Temporary daily hypercapnia for 2 hours between day 4 and 14 after SAH

SUMMARY:
Temporary hypercapnia leads to a reproducible increase of cerebral blood flow (CBF) and brain tissue oxygenation (StiO2) as shown in a previous study (Trial-Identification: NCT01799525). The aim of this study now was to measure the course of carbon dioxide partial pressure (pCO2) reactivity after prolonged hypercapnia, and to evaluate the therapeutic effect of graded hypercapnia.

DETAILED DESCRIPTION:
Cerebral vasospasm still is the leading cause of delayed cerebral ischemia (DCI) and secondary ischemic deficits after aneurysmal subarachnoid hemorrhage (SAH). Hypercapnia leads to a reproducible increase of cerebral blood flow (CBF) and brain tissue oxygenation (StiO2) as shown in a previous study (Trial-Identification: NCT01799525). Furthermore, the increase of CBF and StiO2 sustained after normalization of ventilation and no rebound effect was found. So, a possible optimization of the hypercapnic period may lead to prolonged effects of increased CBF and StiO2. Aim of this stuy is to find the ideal duration of hypercapnia and to evaluate the therapeutic effect of graded hypercapnia. For this, intubated and mechanically ventilated patients with an aneurysmal SAH Hunt/Hess 3-5, Fisher grade 2-4 on the initial CT scan and supplied with an external ventricular drainage will be included within the first 96 hours after ictus. Between day 4 and 14 they undergo a trial intervention in which the respiratory minute volume will be reduced in order to maintain a target PaCO2 of 50 - 55 mmHg for 2 hours. Arterial blood gas analysis (ABG) and transcranial Doppler sonography (TCD) is performed in 15-minute intervals. Intracranial pressure (ICP), cerebral perfusion pressure (CPP), and cardiovascular parameters are monitored continuously, serial measurement of CBF and StiO2 under continous hypercapnia is performed. Primary endpoint of this trial is change of CBF under hypercapnia, secondary endpoints are StiO2, measures non-invasively with near-infrared spectroscopy, mean flow velocity of intracranial vessels in TCD, delayed cerebral infarction in cranial CT and Glasgow Outcome Score (GOS) after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal SAH
* Aneurysm occluded by clipping/coiling within 96 hours
* Hunt/Hess 3-5
* Fisher 2-4 on initial CT scan
* Intubated, sedated and mechanically ventilated patient
* Continous drainage of cerebrospinal fluid (CSF)

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Common obstructive lung disease (COLD)
* potential of hydrogen (pH) in ABG < 7,25
* ICP > 20 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow (CBF) | 2-4 hours, day 4-14 after SAH
  Changes of CBF (absolute, ml/100g tissue/min) under changes of arterial pCO2

SECONDARY OUTCOMES:
Cerebral tissue oxygen saturation | 2-4 hours, day 4-14 after SAH
  Changes of tissue oxygen saturation measured by near-infrared spectroscopy (NIRS)
Glasgow Outcome Score (GOS) | up to 6 months
  Glasgow Outcome Score (GOS 1 - 5, GOS 1 = Death, GOS 5 = none or low disability) after 14 days, after discharge and 6 months

IPD SHARING:
Plan to Share IPD: Undecided